CLINICAL TRIAL: NCT06929390
Title: A Prospective, Multicenter, Randomized Controlled Clinical Trial Comparing Bronchoscopic Thermal Vapor Ablation and Percutaneous Microwave Ablation in Patients With COPD and Early-Stage Lung Cancer: Efficacy and Safety Evaluation
Brief Title: Comparing BTVA and MWA in COPD With Early Lung Cancer: Efficacy and Safety
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henan Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Xiaoju Zhang
Record Dates: First submitted 2025-01-14; First posted 2025-04-16 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Copd; Lung Cancer
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- bronchoscopic thermal vapor ablation (Experimental): Patients will undergo bronchoscopically guided thermal vapor ablation therapy
  Interventions: Procedure: BTVA
- percutaneous microwave ablation (Experimental): Patients will undergo CT-guided percutaneous microwave ablation therapy
  Interventions: Procedure: MWA

INTERVENTIONS:
Procedure: BTVA — The eligible subjects will be stratified according to stratification factors (pure GGN/mixed GGN, lesion size ≤1cm/>1cm, FEV1 ≤50%/>50%) and randomized at a 1:1 ratio to two groups. Patients in the BTVA group will undergo BTVA treatment.
  Arms: bronchoscopic thermal vapor ablation
Procedure: MWA — The eligible subjects will be stratified according to stratification factors (pure GGN/mixed GGN, lesion size ≤1cm/>1cm, FEV1 ≤50%/>50%) and randomized at a 1:1 ratio to two groups. Patients in the MWA group will undergo MWA treatment.
  Arms: percutaneous microwave ablation

SUMMARY:
Based on the advantages of BTVA in the treatment of early-stage lung cancer and COPD, researchers propose the concept of using BTVA to treat COPD combined with early-stage lung cancer. Researchers plan to conduct a multicenter clinical study focusing on patients with COPD combined with malignant GGNs. Bronchoscopic BTVA surgery or percutaneous MWA surgery will be performed, evaluating the effectiveness and safety of bronchoscopic BTVA and percutaneous MWA surgery in the treatment of COPD combined with early-stage lung cancer.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a common respiratory disease, affecting nearly 100 million people in China, with the highest mortality rate globally. It is strongly associated with lung cancer, as both share risk factors such as tobacco exposure and environmental pollution. Additionally, chronic inflammation and abnormal repair mechanisms in COPD further increase the risk of lung cancer. Early diagnosis and treatment of lung cancer are crucial, particularly in detecting pulmonary nodules (GGN). Although malignant GGNs progress slowly, early surgical resection remains the best curative option. However, COPD patients face high surgical risks and should carefully consider their treatment options.

Microwave ablation (MWA) has been widely used as a local treatment for early-stage lung cancer, showing similar efficacy to surgery. However, percutaneous procedures may lead to complications such as pneumothorax and bleeding. In contrast, bronchoscopic thermal vapor ablation (BTVA), performed under general anesthesia, avoids the drawbacks of local anesthesia, enables precise tumor ablation, and improves lung function. Studies suggest that BTVA holds great promise for the treatment of both COPD and lung cancer, offering a new therapeutic option.

Based on the advantages of BTVA in the treatment of early-stage lung cancer and COPD, Researchers propose the concept of using BTVA to treat COPD combined with early-stage lung cancer. Researchers plan to conduct a multicenter clinical study focusing on patients with COPD combined with malignant GGNs. Bronchoscopic BTVA surgery or percutaneous MWA surgery will be performed, evaluating the effectiveness and safety of bronchoscopic BTVA and percutaneous MWA surgery in the treatment of COPD combined with early-stage lung cancer.

ELIGIBILITY:
Inclusion Criteria:

Subjects meeting all of the following criteria are eligible for inclusion:

1. Patients of any gender aged between 35 and 80 years with a diagnosis of chronic obstructive pulmonary disease (COPD);
2. Chest CT showing ground-glass nodules (GGNs) with a solid/tumor ratio (CTR) ≤ 0.25;
3. Nodule size < 2cm located in the upper lobes of both lungs;
4. Pathologically diagnosed as primary peripheral lung cancer, with preoperative clinical staging indicating T1a, bN0M0;
5. Investigator assessment that ablative techniques can be feasibly implemented via bronchoscopic or percutaneous approaches to reach the lesion;
6. Patients unable to undergo surgery or refuse surgery and are unwilling or intolerant to radiation or chemotherapy;
7. Signing an informed consent form, understanding, and actively cooperating with follow-up procedures

Exclusion Criteria:

Subjects meeting any of the following conditions are ineligible for inclusion:

1. Bronchoscopy contraindications, such as:

   1. Myocardial infarction within the past month, unstable myocardial ischemia, ejection fraction (EF) ≤40%
   2. Active hemoptysis
   3. Coagulation disorders
   4. Severe hepatic, renal, cardiac, pulmonary, or cerebral dysfunction, severe anemia, dehydration, and severe nutritional disturbances that cannot be corrected or improved in the short term
2. Pulmonary function reports indicating FEV1 ≤ 20% predicted value, or DLCO ≤ 20%;
3. Respiratory tract infection or acute exacerbation of chronic obstructive pulmonary disease within the preceding 6 weeks before screening;
4. Presence of large bullae in the lobe containing the target lung segment/subsegment (defined as bullae occupying more than 1/3 of the lobe) or paraseptal emphysema;
5. High-density emphysematous changes simultaneously present in the upper and lower lobes of the contralateral lung, defined as HRCT showing low attenuation areas (<-950 HU) comprising more than 40% of the total lung volume;
6. Tumor located within 2cm of the trachea, main bronchi, esophagus, aortic arch branches, main pulmonary artery, left and right pulmonary arteries, or heart, and within 1cm of the nearest pleural boundary;
7. Active pathogenic infection or evidence of active infection (e.g., fever, elevated white cell count), poorly controlled infectious or inflammatory conditions around the lesion or at the puncture site;
8. Discontinuation of anticoagulant and/or antiplatelet medications (excluding new oral anticoagulants such as dabigatran, rivaroxaban) for less than 5-7 days before surgery;
9. Coexisting conditions or medication use increasing the risk of post-treatment complications, including but not limited to: autoimmune disorders, clinically significant immunosuppressants, history of asthma, α-1 antitrypsin deficiency;
10. Daily prednisolone intake exceeding 10mg or an equivalent dose of glucocorticoids during the screening visit;
11. History of cardiac or pulmonary transplantation, surgical lung volume reduction, median sternotomy, endoscopic lung volume reduction (e.g., valves, coils), lobectomy, or lung resection;
12. Eastern Cooperative Oncology Group (ECOG) score >2;
13. Participation in or currently involved in other clinical studies within the past 30 days;
14. Other conditions deemed unsuitable for participation by the investigator.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete ablation rate at 12 months postoperatively | 12 months postoperatively

SECONDARY OUTCOMES:
Technical implementation success rate | On the day of surgery
Complete ablation rate at 6 months postoperatively | 6 months postoperatively
Changes in pulmonary function indicators（FEV1） at 6 months, 12 months, and 24 months post-treatment compared to baseline | 6,12 and 24 months postoperatively
Changes in lung volume assessed by HRCT at 6 months, 12 months, and 24 months post-treatment compared to baseline | 6,12 and 24 months postoperatively
Improvement in exercise tolerance at 6 months, 12 months, and 24 months post-treatment compared to baseline: 6MWD | 6,12 and 24 months postoperatively
Improvement in symptom score（mMRC) at 6 months, 12 months, and 24 months post-treatment compared to baseline | 6,12 and 24 months postoperatively
Local control rates at 1 year, 2 years, and 3 years postoperatively | 1 year, 2 years, and 3 years postoperatively
Progression-free survival (PFS) | 1 year, 2 years, and 3 years postoperatively
Overall survival (OS) | 1 year, 2 years, and 3 years postoperatively
Safety：Evaluate the incidence of (serious) adverse events | On the day of surgery
  Evaluate the incidence of (serious) adverse events related to the device or procedure during the study period.

IPD SHARING:
Plan to Share IPD: No